CLINICAL TRIAL: NCT03972462
Title: Open-label, Fixed-sequence, Two-period Comparative Bioavailability Study of Sirolimus From Topical Application of NPC-12G Gel to Oral Rapamune® Following Single Administration in Healthy Subjects Under Fasting Conditions
Brief Title: NPC-12G Gel 0.2% Sirolimus PK Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: NPC-12G-4/US
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-05

CONDITIONS: Bioavailability Study
MeSH Terms: interventions — Sirolimus; Gels; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NPC-12G Gel 0.2% (Period 1) (Experimental): A single 800 mg quantity weight (1.6 mg sirolimus) dose will be applied to the central face on Day 1.
  Interventions: Drug: NPC-12G Gel 0.2%
- Rapamune Tablet (Period 2) (Active Comparator): Rapamune® (sirolimus) 2 mg tablet for oral dosing.
  Interventions: Drug: Rapamune® 2 mg tablet

INTERVENTIONS:
Drug: NPC-12G Gel 0.2% — Period 1
  Other Names: 2 mg of sirolimus in 1 g of gel
  Arms: NPC-12G Gel 0.2% (Period 1)
Drug: Rapamune® 2 mg tablet — Period 2
  Other Names: Sirolimus
  Arms: Rapamune Tablet (Period 2)

SUMMARY:
This study is designed to describe the relative systemic bioavailability of topical and oral sirolimus formulations.

ELIGIBILITY:
Inclusion Criteria

* Male or female, non-smoker (no use within 3 months prior to screening), ≥ 18 and ≤ 65 years of age, with BMI > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females
* Females of childbearing potential who are sexually active with a male partner must be willing to use one of acceptable contraceptive method throughout the study and for 12 weeks after the last study drug administration

Exclusion Criteria

* Any sign of eczema/dermatitis, skin lesion, wound, or infection at the application site, or any other conditions that would prevent a safe application of the gel formulation.
* Laser or surgery at the gel application site within 2 weeks before the gel application.
* Positive alcohol breath test, urine drug screen or urine cotinine test at screeningation
* History of allergic reactions or hypersensitivity to sirolimus, sirolimus derivatives, or excipient of NPC-12G Gel
* Use of any drugs known to induce or inhibit CYP3A4 metabolism within 30 days prior to the first study drug administration
* Positive pregnancy test at screening
* Breast-feeding subject
* History of active tuberculosis or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening
* Positive QuantiFERON®-TB test with positive chest X-ray, indicating possible tuberculosis infection
* Immunization with a live attenuated vaccine within 1 month prior to dosing or planned vaccination during the study and up to 3 weeks after the last study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
AUC0-48 | Sampling: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose
Cmax | Sampling: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose
Tmax | Sampling: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- InVentiv Health Clinical Research Services LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No